CLINICAL TRIAL: NCT04172519
Title: Evaluation of the Effectiveness of Pelvic Floor Muscles Training for Urinary Incontinence After Radical Prostatectomy. Pilot Study.
Brief Title: Pelvic Floor Muscles Training After Radical Prostatectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Agnieszka Radzimińska, Study Director, Nicolaus Copernicus University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NicolausCU
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Floor Disorders; Urinary Incontinence; Prostatectomy
Keywords: pelvic floor muscles training; laparoscopic radical prostatectomy; adenomectomy
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence | interventions — Lead

STUDY DESIGN:
Intervention Model Description: Parallel crossover study
Who Masked: Participant, Outcomes Assessor
Masking Description: Stratified randomization was ensured by allocating the subjects using a simple method. One person picked envelopes with group allocation numbers from a computer generated random number table. It should be noted that the main investigator was blinded during the group allocation process. The randomized control trials (RCT) reporting quality has been improved using the CONSORT statement (Consolidated Standards of Reporting Trials).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Patients who before prostate cancer surgery will receive: psychological consultation, nursing consultation, physiotherapy consultation and intervention (4 visits which will be implemented pelvic floor muscle training). Then patients will have radical laparoscopic prostatectomy, after which (after 2 and 6 weeks) they receive psychological consultation, nursing consultation (immediately after surgery) and physiotherapeutic consultation (supervised exercises - meeting twice a week with a physiotherapist, after 2 weeks from surgery for 3 months - 24 interventions, patients for three months additionally perform the recommended exercises 3 times a day at home for 3 months on their own). Then, 6 months after the surgery, there will also be a physiotherapy consultation.
  Interventions: Other: Pre- and post prostatectomy supervised PMFT
- Group B (Experimental): Patients who will receive: psychological consultation, nursing consultation, physiotherapy consultation before prostate cancer surgery. Subsequently, patients will have the procedure performed laparoscopic radical prostatectomy, immediately after which they receive psychological consultation, nursing consultation. The physiotherapist consultation will be two weeks after the surgery, during which the physiotherapist will provide an instruction pelvic floor muscle training. Patients do the exercises themselves at home according to the instructions, 3 times a day for 3 months). Physiotherapeutic consultation 6 months after surgery.
  Interventions: Other: Unsupervised PMFT
- Group C (Experimental): Patients who will not receive any intervention before prostate cancer surgery. Then patients will have radical laparoscopic prostatectomy, after which (after 2 and 6 weeks) they receive psychological consultation, nursing consultation (immediately after surgery) and physiotherapeutic consultation (supervised exercises - meeting twice a week with a physiotherapist, after 2 weeks from surgery for 3 months - 24 interventions, patients for three months additionally perform the recommended exercises 3 times a day at home for 3 months on their own). Physiotherapeutic consultation 6 months after surgery.
  Interventions: Other: Supervised PMFT
- Group D (No Intervention): Control group, patients after radical laparoscopic prostatectomy, without additional interventions

INTERVENTIONS:
Other: Pre- and post prostatectomy supervised PMFT — intervention before and after surgery, supervised exercises
  Arms: Group A
Other: Unsupervised PMFT — intervention after surgery, unsupervised exercises
  Arms: Group B
Other: Supervised PMFT — intervention after surgery and supervised exercise
  Arms: Group C

SUMMARY:
Prostate cancer (PCa) is a malignant tumor commonly diagnosed among men in the USA and Europe. About 81% of cases of prostate cancer are detected early on, which allows patients to receive effective treatment. High risk cancer patients may undergo radical prostatectomy (RP) which includes the removal of the entire prostate gland together with both seminal vesicles, prostatic urethra, and bilateral pelvic lymph nodes. Even though RP has been improved over decades, patients are still at risk of surgical and post-surgical complications. The most common complications include urinary incontinence and erectile dysfunction. Pelvic floor muscle training is recognized as the physiotherapeutic modality for the treatment of urinary incontinence in men after radical prostatectomy. This method is recommended by the European Association of Urology. However, the literature analysis and systematic review carried out by our team prove that there are relatively few clinical trials with a well-developed research protocol assessing this form of therapy. In order to objectify the effects of therapy, we will assess both psychosocial aspects, as well as try to answer the question whether biochemical parameters can be a marker of pelvic floor muscles. In previous own research, we obtained promising results by examining biochemical parameters during pelvic floor muscle activity in women with stress urinary incontinence.

DETAILED DESCRIPTION:
The subject of the study is to assess the impact of physiotherapeutic intervention in the form of pelvic floor muscle training in patients after laparoscopic radical prostatectomy. A randomized control trials will be carried out on a group of about 300 people (men over 40 years of age) before and after radical prostatectomy. The examined people will be divided into 4 groups and will be assessed before and after surgery: 2 weeks, 6 weeks, 3 months and 6 months. All participants in the study will undergo tests such as: urodynamic, biochemical, MRI, standardized questionnaires regarding the quality of life, physiotherapeutic assessment, histopathological assessment, and cancer progression assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with prostate cancer qualified for surgery
* patients who underwent radical prostatectomy
* 40-85 years of age.
* patients who gave their written consent to participate in the study
* patient's joining the program will always be preceded by a medical consultation and exclusion of contraindications to therapy
* patients able to understand Polish.

Exclusion Criteria:

* classical retropubic operation,
* classical perineal surgery,
* operation assisted by daVinci robot,
* partial prostate surgery,
* transurethral resection of the prostate (TURP),
* the research will not involve incapacitated persons, soldiers of the basic service, persons deprived of their liberty and remaining in official or other dependence with the persons conducting the examination,
* patient's disagreement to participate in pelvic floor muscle training
* intraoperative and postoperative complications preventing the introduction of early rehabilitation ((damage to the external sphincter, urinary tract infection, bladder neck narrowing),
* prostate cancer recurrence,
* no incontinence after surgery,
* urinary incontinence before surgery,
* previous prostate surgery.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
General Self Efficacy Scale (GSES) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  The raw scores are afterward transformed into standardized sten scores. The higher the score, the higher are self-efficacy beliefs. Score ranges are defined as follows: 1-4 sten, low scores; 5-6 sten, average scores; and 7-10 sten, high scores.
Self Esteem Scale (SES) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  General Self-Assessment Level Scale is a tool that allows you to assess the level of general self-assessment. It consists of 10 diagnostic statements. The test is designed to indicate the four-level scale, to what extent patients agree with each of these statements. The raw results obtained are converted into standardized sten standards. The following scoring is taken: 1-4 sten - low results; 5-6 sten - average results; 7-10 sten - high results.
Beck Depression Inventory - II (BDI - II) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  The BDI questionnaire has been the most widely used self-report depression scale. The tool is used in research on mental disorders and to assess the mood of patients suffering from various medical conditions, including oncological, urological, gynecological, and neurological diseases. The BDI-II questionnaire is a 21-item scale with individual item scores ranging from 0 (no symptoms) to 3 (severe symptoms). A total score of 0-8 is considered as no depression, 9-18 indicates moderate depression, and a score of 18+ is considered as severe depression.
Acceptance of Disease Scale (AIS) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Acceptance of Disease Scale (AIS) which determines the extent to which the patient accepts his own illness and assesses the severity of negative emotions associated with it. This tool contains 8 statements describing the consequences of the disease. Each statement is scored 1-5 (1- lack of acceptance of the disease; 2-5 good adaptation to the disease situation).
International Index of Erectile Function - 5 (IIEF - 5) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  The International Index of Erectile Function - 5, which consists of 15 items and 5 domains, is a psychometrically valid and reliable instrument that was developed through consultations with an international panel of experts for use in determining efficacy of treatment in controlled clinical trials.
Expanded Prostate Cancer Index Composite-26 (EPIC-26) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  EPIC-26, contains five symptom domains (urinary incontinence, urinary irritative/obstructive, sexual, bowel, hormonal), scored from 0 (worst) to 100 (best), that can be tracked over time to understand symptom burden, functional outcomes and the impact of side effect management strategies.
EORTC Quality of life Questionnaire -Prostate Cancer Module (EORTC QLQ-PR25) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  The prostate-specific module EORTC QLQ-PR25 is a self-administered questionnaire that includes 4 subscales for assessment of Urinary symptoms (9 items, labeled US31-US39), Bowel symptoms (4 items, BS40-BS43), Hormonal treatment-related symptoms (6 items, TS44-TS49), and Sexual activity and function (6 items, SX50-SX55).
EORTC Quality of Life Questionnaire core 30 (EORTC QLQ-C30) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  EORTC QLQ-C30 assesses HRQoL in cancer patients with 15 scales, each ranging in scores from 0 to 100.
International Prostate Symptom Score (I-PSS) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Sex Hormone Binding Globulin (SHGB) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
Luteinizing Hormone (LH) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
Follicle Stimulating Hormone (FSH) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
Free testosterone | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  The test is performed in cases where the interpretation of total testosterone results is questionable or impossible due to fluctuations in SHBG levels.
Total testosterone | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
Colecalciferol (vitamin D3.) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  In the blood should be in the range of 30-50 nmol / l (20 ng / ml).
Myostatin | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting into Vacuette tubes with EDTA anticoagulant. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
Irisin | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Six milliliters of blood will be collected from each subject after at least 12 hours fasting into Vacuette tubes with EDTA anticoagulant. Participants had to fast over night with the last meal before 7 pm on the day before the investigation.
N-terminal telopeptide of type 1 collagen (NTX) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Morning urine collection
C-telopeptide of type 1 collagen (CTX) | 1 day 2 weeks before surgery and assessment of change from baseline at 6 weeks, 3 months and 6 months after operation
  Morning urine collection
Multi-parametric pelvic magnetic resonance (mp NMR) | 2 days
  with evaluation of the prostate gland before surgery and lodge of prostate gland after radical prostatectomy
Gleason Score | 1 day
  The Gleason Score ranges from 1-5 and describes how much the cancer from a biopsy looks like healthy tissue (lower score) or abnormal tissue (higher score). Most cancers score a grade of 3 or higher.
Histopathological examination questionnaire | 1 day
  operator's assessment
TNM Classification of Malignant Tumors (TNM) | 1 day
  Small, low-grade cancer, no metastasis, no spread to regional lymph nodes, cancer completely removed, resection material seen by pathologist: pT1 pN0 M0 R0 G1; this grouping of T, N, and M would be considered Stage I.
  Large, high grade cancer, with spread to regional lymph nodes and other organs, not completely removed, seen by pathologist: pT4 pN2 M1 R1 G3; this grouping of T, N, and M would be considered Stage IV.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Radzimińska, PhD, Study Director — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Aleksander Goch, Prof., Study Chair — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Katarzyna Strojek, PhD, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Magdalena Weber-Rajek, PhD, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Agnieszka Strączyńska, PhD, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Zuzanna Piekorz, PhD, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Hanna Styczyńska, PhD, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz; Piotr Jarzemski, MD, PhD, Study Director — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz,; Stanisław Wroński, MD, PhD, Principal Investigator — The Jan Biziel Hospital in Bydgoszcz, Department of Urology; Piotr Słupski, MD, Principal Investigator — The Jan Biziel Hospital in Bydgoszcz, Department of Urology; Beata Pilasrka, RN, Principal Investigator — Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz,; Marcin Jarzemski, MD, Principal Investigator — The Jan Biziel Hospital in Bydgoszcz, Department of Urology; Bartosz Brzoszczyk, MD, Principal Investigator — The Jan Biziel Hospital in Bydgoszcz, Department of Urology
Locations (2):
- Poland (2):
  - The Jan Biziel Hospital, Department of Urology, Bydgoszcz
  - Nicolaus Copernicus University in Torun Collegium Medicum in Bydgoszcz, Department of Physiotherapy, Bydgoszcz

IPD SHARING:
Plan to Share IPD: No
Individual participant data, can be available at the request of interested parties.